CLINICAL TRIAL: NCT06541795
Title: Evaluation of Long-term Safety and Performance of AcrySof IQ Vivity Extended Vision and AcrySof IQ Vivity Toric Extended Vision Intraocular Lenses
Brief Title: Evaluation of AcrySof IQ Vivity Extended Vision Intraocular Lenses
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Management decision
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILI875-I001
Record Dates: First submitted 2024-08-01; First posted 2024-08-07 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Aphakia; Presbyopia; Residual Refractive Cylinder
Keywords: Cataracts
MeSH Terms: conditions — Aphakia; Presbyopia; Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- AcrySof IQ Vivity Extended Vision IOL and AcrySof IQ Vivity Toric Extended Vision IOL (Experimental): AcrySof IQ Vivity Extended Vision IOL implanted in both eyes during cataract surgery
  Interventions: Device: AcrySof IQ Vivity Extended Vision IOL

INTERVENTIONS:
Device: AcrySof IQ Vivity Extended Vision IOL — UV-absorbing, with or without blue light filtering, foldable IOL implanted in the capsular bag of the eye for the visual correction of aphakia in adult patients from whom a cataractous lens has been removed. The IOL mitigates the effects of presbyopia by providing an extended depth of focus. The toric models in addition reduce residual refractive astigmatism in patients with pre-existing corneal astigmatism.
  Other Names: AcrySof IQ Vivity Extended Vision IOL: Model DFT015; AcrySof IQ Vivity Extended Vision UV Absorbing IOL: Model DAT015; AcrySof IQ Vivity Toric Extended Vision IOL: Models DFT215, DFT315, DFT415, DFT515 and DFT615 according to country of conduct; AcrySof IQ Vivity Toric Extended Vision UV Absorbing IOL: Models DAT315, DAT415, DAT515 and DAT615 according to country of conduct

SUMMARY:
The purpose of this post-market study is to describe the long-term safety and performance of AcrySof IQ Vivity and AcrySof IQ Vivity Toric intraocular lens (IOL) models in a real-world setting through routine clinical practice.

DETAILED DESCRIPTION:
This study includes a retrospective chart review to obtain preoperative, operative, and post-operative data, and one prospective visit to collect key long-term safety and performance endpoints in a sample of subjects commercially implanted with the specified IOLs for 3 to 5 years in the real world.

This study will be conducted in the US and in Spain.

ELIGIBILITY:
Key Inclusion Criteria:

* 22 years old or older at Visit 1.
* Able to understand and sign an approved informed consent form.
* Implantation of AcrySof IQ Vivity and/or Vivity Toric IOL models in both eyes for 3 to 5 years prior to enrollment.
* Documented medical history and required pre-operative baseline information available for retrospective data collection.
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria:

* Corneal refractive surgery after AcrySof Vivity or AcrySof Vivity Toric IOL implantation.
* Pregnant or nursing at the time of enrollment.
* Childbirth after IOL implantation.
* Other protocol-specified exclusion criteria may apply.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Mean Binocular Best Corrected Distance Visual Acuity (BCDVA) at Visit 1 | Visit 1, Year 3-5 postoperative
  Visual acuity (VA) will be assessed binocularly (both eyes together) with correction in place using letter charts at a distance of 4 meters. BCVA will be recorded in logarithm Minimum Angle of Resolution (logMAR) LogMAR values typically range from -0.3 (20/10 vision on the Snellen chart) to 1 (20/200 vision). A logMAR acuity of 0.0 corresponds to 20/20 Snellen acuity (normal distance visual acuity), with a negative value denoting better than 20/20 visual acuity. No hypothesis testing is prespecified for this endpoint.
Incidence of adverse events | Up to Year 3-5 postoperative
  An adverse event (AE) is defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users, or other persons, whether or not related to the study device. Adverse events reported or observed since the time of initial exposure to the study model IOL will be recorded.
Incidence of device deficiencies | Up to Year 3-5 postoperative
  A device deficiency is defined as an inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety, or performance. Device deficiencies reported or observed since the time of initial exposure to the study model IOL will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management Operations, Surgical, Study Director — Alcon Research, LLC
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States